CLINICAL TRIAL: NCT02768103
Title: Evaluating Neural Adaptation After Tendon Transfer and Task-based Training in SCI
Brief Title: Neural Adaptation After Tendon Transfer and Training in Tetraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: N1772-P
Record Dates: First submitted 2016-05-06; First posted 2016-05-11 (Estimated); Results first posted 2020-04-15 (Actual); Last update posted 2022-11-15 (Actual); Status verified 2022-10

CONDITIONS: Spinal Cord Injury
Keywords: upper extremity; spinal cord injury; surgical reconstruction; MRI, functional; rehabilitation
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Intervention Model Description: All participants complete 10 week task based training in home setting.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- SCI transfer + training (Experimental): Individuals with tetraplegia and brachioradialis to flexor pollicis longus transfer will participate in 10 week home training program to improve surgical outcome (pinch strength)
  Interventions: Behavioral: task-based training

INTERVENTIONS:
Behavioral: task-based training — The 10-week training program is designed to incorporate requirements of motor learning and includes activities that require learning to coordinate the transferred Br with other synergists by producing pinch force in different upper limb postures and in a range of pinch openings. Biofeedback using a pinch dynamometer in self-selected postures provides feedback and knowledge of progress to the participant. A task board is used for practicing task-specific activities such as opening and closing zippers, using a remote, an ATM card, a key, and an electrical plug and focuses on pinch in dynamic conditions that require modulating force and maintaining specific positions. The pinch-pin device requires closing pinch-pins (clothes pin) of variable resistance ranging from approximately 1 to 8 lbs and placing them on rods arranged at different positions in the work space.

SUMMARY:
The number of people in the United States who have survived SCI is estimated to be approximately 273,000 persons. Around 50% of the injuries are to the cervical spine resulting in tetraplegia. An important rehabilitation goal in this population is recovery of upper limb function, which could decrease medical costs and improve their quality of life. Re-establishing active grasp and pinch strength to the hand can be accomplished by surgeries that transfer the tendon of a strong muscle to restore strength to a paralyzed muscle, but the outcomes of the surgeries are variable. The investigators have demonstrated in an ongoing study, the functional gains after surgery can be improved with a focused therapy program to retrain the transferred muscle. The propose of this study is to examine the cortical mechanisms that drive successful muscle re-education after surgery. Understanding the neural (brain) activity associated with functional performance can help to predict who will respond to therapy and will guide evidence-based rehabilitation programs to improve upper limb function in tetraplegia.

DETAILED DESCRIPTION:
Restoring upper limb function is rated among the highest priorities for individuals with tetraplegia. Re-establishing active grasp and pinch strength to the hand can be accomplished by tendon transfer procedures in which the tendon of a strong proximal muscle is surgically re-attached to the tendon of a paralyzed muscle. A common procedure to restore lateral (key) pinch is to transfer the distal tendon of one of the three elbow flexor muscles, the brachioradialis (Br) to the tendon of the paralyzed thumb flexor, the flexor pollicis longus (FPL). Recovery of functional pinch depends on how well the patient learns to activate the Br to flex the thumb through its new distal attachment, and also to control flexion at the elbow through its proximal attachment. The investigators' previous work shows that Br to FPL recipients do not activate the transferred Br fully and may not reach optimal functional status on their own or with traditional therapies. The investigators propose that participation in a postoperative task-based training program will drive cortical changes that impact functional (pinch) ability.

Recent studies of individuals with cervical SCI show substantial cortical reorganization can occur after the injury, but neural substrates of motor learning after tendon transfer have not been studied. For these patients, very little is known about what functional brain changes accompany improved performance in response to additional intervention. The Br to FPL transfer alters the central feedback from the periphery and may permit new or adaptive neural pathways that can achieve greater functional use of the tendon transfer. Neuroimaging techniques, such as functional magnetic resonance imaging (fMRI) have become important tools for understanding plasticity in the neuromuscular system and for assessing the neural underpinnings of successful novel interventions. The objective of the proposed study is to identify the neural pattern that is associated with the best functional outcomes (highest pinch force) after Br to FPL transfer. The investigators will use fMRI and functional performance measures to find neural predictors and correlates of muscle re-education. That is, the investigators expect that successful postoperative muscle re-education will depend on increased cortical drive to the transferred Br in combination with new synergists, and this will be reflected in the neural imaging results.

The purpose of the study is to evaluate neural activity from Br to FPL transfer recipients after conventional therapy and in response to an additional task-based training home program that aims to improve voluntary activation of the transferred Br in functional pinch tasks. The 10-week training program is under evaluation in RRD Pilot (B0583P) study and includes producing pinch force in different upper limb postures, biofeedback from a pinch dynamometer, and practicing selected pinch tasks. The investigators anticipate that increases in the amplitude and distribution of fMRI blood oxygen level dependent (BOLD) responses in sensorimotor cortices will underlie improved motor control post-surgically and following successful intervention to promote motor relearning.

Specific Aims

1. Define the cortical representation of pre-training pinch function in SCI patients. The investigators will quantify the pattern (location, volume and intensity) of cortical activation associated with voluntary pinch in individuals who are one-year post Br to FPL tendon transfer surgery and a conventional therapy program. The investigators hypothesize (H1) greater volume and intensity of brain activation will correlate to better pinch function measured by pinch strength and the magnitude Br activation in pinch. Secondary analyses will determine if the location of the brain activation varies with pinch function (force) and specificity relative to voluntary elbow flexion.
2. Evaluate the cortical response to the task-based home therapy program. Correlates of task-based adaptation from pre- to post-training will be assessed using fMRI. H2: Greater activation (intensity and volume) in the primary motor cortex (M1) and sensory cortex will translate to increased voluntary activation of the transferred Br in pinch compared to elbow flexion. Task-based training outcome measures will include isometric pinch force magnitude, EMG quantification of Br activation in pinch and elbow flexion.
3. Determine neural signatures of surgical and training induced motor improvements. H3: After directed task-based training, brain activity during voluntary pinch will extend to adjacent areas (larger representation, greater activity), in sensorimotor brain areas, facilitating the ability to voluntarily increase the transferred Br activation in pinch. Secondary analyses will contrast size and activation level of brain changes with pinch activation in patients who receive training relative to non-impaired and non-surgical participants.

The postoperative therapy protocols after tendon transfer procedures are not well defined, inconsistently applied, and lack evidence for their effectiveness. The study proposed here will investigate cortical change to assess outcome dependent plasticity. Thus, it may be possible to predict why some individuals do not re-train the transferred muscle as well as others. Establishing this relationship can lead to understanding the mechanisms of successful interventions and may identify brain based dynamics that could become the focus of future treatments (e.g. biofeedback, brain stimulation, etc.).

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a clinical diagnosis of SCI cervical level 4-7, complete or incomplete injuries, who have completed conventional therapy and be at least 1-year post-surgery, are eligible for the study.
* Participants must have had Br to FPL tendon transfer, be willing to participate in a 10 week exercise program, have adequate assistance or be independent in setting up exercise equipment (weight cuffs, functional tasks), and be available for two measurement sessions.
* Women and minorities may be included in the study if they meet the inclusion criteria.
* Non-Veteran participants who meet the selection criteria will be included to expand the available number of subjects.

Exclusion Criteria:

* More than one tendon transfer to the thumb to restore pinch but not if they have other tendon transfer procedures on the same upper limb.
* Other exclusion criteria include pain that would limit their ability to perform the activities, spasticity in the upper limb, or spinal cord injury level above C4 or below C7 as their pattern of weakness will be substantially different.
* Subjects who are participating in other research studies that include exercise programs for the upper limb or drug studies that affect their response to exercise will also be excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mary E Johanson, DPT, Principal Investigator — VA Palo Alto Health Care System, Palo Alto, CA
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, CA, Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Johanson ME, Dairaghi CA, Hentz VR. Evaluation of a Task-Based Intervention After Tendon Transfer to Restore Lateral Pinch. Arch Phys Med Rehabil. 2016 Jun;97(6 Suppl):S144-53. doi: 10.1016/j.apmr.2015.12.032. PMID 27233589

RESULTS

PARTICIPANT FLOW:
Groups:
- SCI Transfer + Training: Individuals with tetraplegia and brachioradialis to flexor pollicis longus transfer will participate in 10 week home training program to improve surgical outcome (pinch strength)
  task-based training: 10-week training program incorporates activities that require learning to coordinate the transferred Br with other synergists by producing pinch force in different upper limb postures and in a range of pinch openings. Biofeedback using a pinch dynamometer in self-selected postures provides feedback to the participant. A task board is used for practicing task-specific activities such as opening and closing zippers, using a remote, an ATM card, a key, and an electrical plug and focuses on pinch in dynamic conditions that require modulating force and maintaining specific positions. The pinch-pin device requires closing pinch-pins (clothes pin) of variable resistance ranging from approximately 1 to 8 lbs and placing them on rods arranged at different positions in the work space.
Period: Overall Study
Arm/Group | SCI Transfer + Training
Started | 5
Completed | 4
Not Completed | 1
Not completed — 1 participant did not fit in the fMRI | 1

BASELINE CHARACTERISTICS:
Arm/Group | SCI Transfer + Training
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 4
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Pinch force [Mean (Standard Deviation); unit: Newtons] | 8.7 (6.5)

OUTCOME MEASURES:

1. Primary Outcome: Pinch Force
Description: Pinch force recorded in newtons from force sensor mounted to a custom grip
Time Frame: after 10 weeks home exercise program with task-based training
Measure: Mean (Standard Deviation); unit: newtons
Arm/Group | SCI Transfer + Training
Number analyzed (Participants) | 4
newtons
  Pre-training pinch force (N) | 8.7 (6.5)
  Post-training pinch force (N) | 10.6 (8.6)

2. Primary Outcome: Functional MRI BOLD Signal From Motor Cortex
Description: A block design with 10 seconds of rest alternating with 10 seconds of functional movement for 6 minutes will be followed. Participants have visual cues to instruct them in the timing and sequence of the tasks to be performed. Scan time to include a session of elbow flexion and a session for pinch is about 20 minutes. The main outcome measures for the fMRI data will be brain activation defined by intensity and cluster size in response to performing elbow flexion and pinch. Second level analyses will be mixed models effects derived using FSL FLAME for within subjects (pre to post intervention) as well as cross-sectional (non impaired vs. SCI-ns; SCI-ns vs. SCI+TT) individual models (with outlier deweighting and standard settings).
Time Frame: after 10 week home exercise program with task-based training
Population: No valid data were recorded. The fMRI data collection program had errors in the protocol that rendered the data useless.
Arm/Group | SCI Transfer + Training
Number analyzed (Participants) | 0

3. Secondary Outcome: Fine-wire Electromyography of Transferred Brachioradialis Muscle (to Paralyzed Thumb Flexor)
Description: EMG signal recorded from fine-wire (intramuscular) electrodes normalized to a maximum voluntary contraction
Time Frame: after 10 week home exercise program with task-based training
Measure: Mean (Standard Deviation); unit: percentage of Max Br Contraction
Arm/Group | SCI Transfer + Training
Number analyzed (Participants) | 4
percentage of Max Br Contraction
  pre-training normalized Br EMG | 30 (10)
  post training normalized Br EMG | 34 (10)

ADVERSE EVENTS:
Time Frame: Adverse event data were collected during the 10 week training period.
Groups:
- SCI Transfer + Training: Individuals with tetraplegia and brachioradialis to flexor pollicis longus transfer participate in 10 week home training program to improve surgical outcome (pinch strength). The 10-week training program includes activities that require learning to coordinate the transferred Br with other synergists by producing pinch force in different upper limb postures and in a range of pinch openings. Biofeedback using a pinch dynamometer in self-selected postures provides feedback and knowledge of progress to the participant. A task board is used for practicing task-specific activities such as opening and closing zippers, using a remote, an ATM card, a key, and an electrical plug and focuses on pinch in dynamic conditions that require modulating force and maintaining specific positions. The pinch-pin device requires closing pinch-pins (clothes pin) of variable resistance ranging from approximately 1 to 8 lbs and placing them on rods arranged at different positions in the work space.
Arm/Group | SCI Transfer + Training
All-Cause Mortality (participants affected / at risk) | 0/4
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
No valid data to report for functional MRI outcome.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-31): https://cdn.clinicaltrials.gov/large-docs/03/NCT02768103/Prot_SAP_000.pdf